CLINICAL TRIAL: NCT06921018
Title: Bioavailability of Micronutrients With a Special Focus on Vitamin K - Study Part II: PLANTEKOST
Brief Title: Bioavailability of Micronutrients With a Special Focus on Vitamin K Dependent on Consumed Diet
Acronym: BioMicro
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Technical University of Denmark (Other)
Responsible Party: Principal Investigator, Susanne Bügel, Professor, Head of Section, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: BioMicro Prot. v1.1 PLANTEKOST
Record Dates: First submitted 2025-03-12; First posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Micronutrient Status
Keywords: Bioavailability; Micronutrients; Vitamin K; vitamin B2; Vitamin B12; zinc; iodine; haemoglobin
MeSH Terms: interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vegan diet (Experimental): The participants will consume a vegan diet
  Interventions: Behavioral: change in diet
- average habitual danish diet with high meat consumption (No Intervention): average habitual danish diet with high meat consumption

INTERVENTIONS:
Behavioral: change in diet — the participants will either be assigned consumption of a vegan diet or their habitual average danish diet with a high intake of meat for the intervention period which is 4 weeks.
  Other Names: diet
  Arms: Vegan diet

SUMMARY:
Objectives

The main objectives are:

• Study part II: to investigate the effect of a plant-based diet on micronutrient status compared to an average Danish diet

Hypotheses Study part II: it is hypothesised that the status of some micronutrients is lower after intake of a plant-based diet compared to an average Danish diet.

Participants will:

Study part II: consume either a vegan diet or an average danish diet with a high meat intake for 4 weeks. The total study period for the participants is estimated to 6 weeks (from screening to paticipants last visit)

DETAILED DESCRIPTION:
Overall study design Study part II (n= 16 completers): A 4-week randomised parallel intervention trial comparing status of some micronutrients (with main focus on MK-9 and ferritin) after consumption of a plant-based diet compared to an average Danish diet

In study part II, participants will be randomised to either plant-based or an average Danish (meat-based) diet for 4-weeks. The participants will visit NEXS for two test days, before and after the 4-week intervention period where fasting blood will be drawn. Prior to the two test days the participants will complete a 3-day weighed dietary registration (WDR) and collect faecal and urine samples. The minimum duration for each participant will be 33days.

It is required that the participants' vitamin D status is stable. Therefore, a run-in period of up to 6-week with daily supplementation of vitamin D will be required before the first test day.

Detailed study design of part II Prerequisites Six weeks before the first test day it is required that participants have been supplemented with 10 µg vitamin D3/day (recommended daily intake) and restrain from all other types of (vitamins and mineral) supplementation. The vitamin D supplements will be provided free of charge. On day -5 (or at screening) the participants will show up at NEXS where they will receive containers and cooler bags for urine and faecal sampling. The participants will further get written and oral instructions for the WDR. Prior to Day 0, the participants will perform a 3-day WDR, collect a spot faecal sample and a 24-hour urine sample. Prior to the test day, alcohol is prohibited 48 hours before, high-intensity physical activity is prohibited 24 hours before and the participants will fast for a minimum of 12 hours before. The participants are allowed to drink ½ L of tap water during the fasting period.

Test days On Day 0, the participants will show up fasting at NEXS and one fasting blood sample will be collected (baseline blood sample). The participants will have a session with a dietician, or other delegated personnel, where they will be introduced to their assigned diets (both including daily supplementation with 10 µg vitamin D3) and asked to start the 4-week intervention. On Day 28 (±3 days), the participants will have their second test day at NEXS where one blood sample will be drawn. Prior to the second test days (Day28), they repeat the 3-day WDR, sampling of faeces and urine, and prerequisites related to alcohol intake, physical activity and fasting is required as described above.

Intervention period During the 4 weeks, the participants will show up at NEXS 1-2 days per week to receive new products and if needed they can ask for recipes, guidelines and feedback/advice from a trained dietician. Once a week they will be asked to collect a spot urine sample in the morning on the day they visit NEXS. During the third week, participants will in addition to the above mentioned also have instructions for the WDR and collections of urine and faeces repeated, and material delivered.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* Between 18 and 65 years old (including both 18 and 65 year olds)
* Danish-speaking
* Willingness to consume/comply with consumption of study-related intervention products/diet
* Willing to take 10 µg vitamin D3/day and omit intake of all other (vitamins and mineral) supplements before and during the trial
* BMI ≤ 30.0 kg/m2
* Habitual consumption of meat at dinner minimum 5 times per week. Meat is defined as red meat and poultry, where red meat is consumed at dinner at least 2 out of 5 times per week (fish consumption is not included in the "5 per week" meat definition).

Exclusion Criteria:

* Daily smokers/users of all kinds of nicotine-containing products.
* Occasional smokers/user can be included if they are willing to refrain from all kinds of nicotine-containing products during the trial (from screening to end of trial)
* Blood donation <3 months prior to study-related blood sampling
* Intensive physical training (> 10 hours of strenuous physical activity per week)
* Participation in other clinical studies at the time of the study
* Pregnant, lactating or planning to become pregnant within the study period
* Habitual alcohol intake above current recommendation (> 10 alcoholic units/week)
* History of cancer within the past five (5) years except basal cell skin cancer and cervix
* Diagnosed with chronic inflammation disorders
* Diagnosed with gastrointestinal diseases
* Diagnosed with bone related diseases
* Diagnosed with psychiatric disorder including depression that requires medical treatment
* Medical treatment of diabetes
* Medical treatment of cardiovascular related disease
* Surgical change of the gastrointestinal tract (removal of appendix is allowed)
* Use of prescription medication that can affect their safety or impact on data
* Inability, physically or mental, to comply with the procedure required by the study protocol and evaluated by the principal investigator (PI), study manager or clinical responsible

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2031-06-30 (Estimated)

PRIMARY OUTCOMES:
Differences in the status of micronutrients dependent on consumption of either a plant-based diet or an average Danish diet | From screening the last visit of the participant will take place after 10 weeks.
  The status of the micronutrients will be assesed by analysing blood, feases and urine samples for biomarkers and concentration of the micronutrients.
  For vitamin K, we will measure the concentration of vitamin K vitamers in blood, feaces and urine and the concentration of the biomarkers MGP and OC in the blood samples.

CONTACTS AND LOCATIONS:
Overall Officials: Susanne G Bügel, Professor, Principal Investigator — University of Copenhagen
Locations (1):
- University of Copenhagen, Frederiksberg, Denmark

IPD SHARING:
Plan to Share IPD: No
We will report anonymized data for publications of the result.